CLINICAL TRIAL: NCT03591458
Title: The Use of Amitriptyline for Improving Hypoglycemia Course and Recognition
Brief Title: Amitriptyline in Treating Hypoglycemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow subject enrollment, unable to complete trial in a timely manner
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB_00110853
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Type1 Diabetes Mellitus; Hypoglycemia Unawareness
MeSH Terms: interventions — Amitriptyline

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amitriptyline (Experimental): Participants will be initiated on 25 mg Amitriptyline daily for two weeks during the Titration Period. Amitriptyline dose will be increased to 50 mg daily for 8 weeks during the Intervention Period. Finally, the dose of Amitriptyline will be reduced to 25 mg daily during the two week Taper Period.
  Interventions: Drug: Amitriptyline
- Placebo (Placebo Comparator): Participants will be initiated on a daily Placebo capsule matching the 25 mg Amitriptyline during the Titration Period. The daily dose will be changed to the Placebo capsule matching the 50 mg Amitriptyline for 8 weeks during the Intervention Period. Finally, the daily dose will be changed back to the Placebo capsule matching the 25 mg Amitriptyline during the two week Taper period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Participants will receive a supply of Amitriptyline capsules for titration, intervention, and taper periods.
  Arms: Amitriptyline
Drug: Placebo — Participants will receive a supply of Placebo capsules, matching those of Amitriptyline, for the titration, intervention, and taper periods
  Arms: Placebo

SUMMARY:
Patients with type 1 diabetes mellitus (T1DM) commonly experience hypoglycemia and develop impaired awareness of hypoglycemia. Many patients using continuous glucose monitoring (CGM) system to mitigate these complications, but continue to spend a significant amount of time in hypoglycemia. The long-term goal is to develop novel and readily available therapeutic approaches to improve hypoglycemia course and awareness in T1DM patients. The objective of this study is to determine whether amitriptyline will improve hypoglycemia course and the ability to recognize hypoglycemic events in T1DM patients who are using CGM.

DETAILED DESCRIPTION:
Poorly controlled T1DM can lead to serious and devastating complications, including microvascular (retinopathy, neuropathy and nephropathy) and cardiovascular disease. Both diabetic microvascular and cardiovascular complications can be reduced by intensive insulin therapy and strict blood glucose aiming for hemoglobin A1C (HbA1c) less or equal to 7%. However, a tighter glycemic control correlates with a higher incidence of hypoglycemia and severe hypoglycemia. As well, recurrent episodes of hypoglycemia reduce patients' ability to recognize hypoglycemic episodes (a condition termed impaired awareness of hypoglycemia). Impaired awareness of hypoglycemia is also associated with an increased risk of severe hypoglycemia. Severe hypoglycemia can lead to seizures, emergency room visits/hospitalization, fear of hypoglycemia, compromised quality of life and potentially death. Thus, hypoglycemia and impaired awareness of hypoglycemia are major barriers to optimal glycemic control.

Real-time continuous glucose monitoring (rtCGM) is a technique which measures interstitial glucose levels every five minutes to estimate coincidental blood glucose levels. A rtCGM will alert patients of hyper/hypoglycemic events at seg glucose thresholds and when the blood glucose levels are rapidly rising/declining. However, many patients using rtCGM continue to have impaired awareness of hypoglycemia and spend a significant amount of time in hypoglycemia.

In an animal model, amitriptyline, a tricyclic antidepressant, demonstrated its ability to completely restore hypoglycemia awareness. This potential effect of amitriptyline on human, however, has not been tested.

In the current study, amitriptyline will be studied as an adjuvant treatment of rtCGM to further improve hypoglycemia course and T1DM patients' ability to recognize hypoglycemic episode.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 Diabetes Mellitus for at least 5 years or more
* Age between 21 to 60 years old
* HbA1c less or equal to 9% with the latest measurement within the last 3 months
* Use of real time Continuous Glucose Monitoring (rtCGM) providing continuous glucose data points for at least 3 months, and at least 80% of CGM readings available over the last 2-week period
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Ongoing or recent history of major depressive disorder, or other ongoing major psychiatric disorders
* History of anti-depressant use within the last three months
* Insulin pump linked to a CGM with programmed automatic insulin adjustment or suspension
* History of advanced cardiac, liver, kidney or neurological disease
* Active malignancy
* Uncontrolled Human Immunodeficiency Virus diseases
* Advanced diabetic retinopathy, neuropathy, or nephropathy
* Frequent acetaminophen use which can disrupt CGM accuracy
* Pregnancy or female of child-bearing potential unable to practice effective contraception during the study period
* Breastfeeding female, or female with prospective plan to initiate breastfeeding
* Ongoing history of alcohol abuse
* Contraindication to amitriptyline use, including hypersensitivity to amitriptyline or any component of the formulation, co-administration with or within 14 days of Monoamine Oxidase Inhibitors and co-administration with cisapride
* Inability to understand or cooperate with study procedures, including taking study drugs and recording hypoglycemic symptoms.

The participants meeting the above criteria will enter "Run-in Period". At the Visit 2, the following additional exclusion criteria will be applied before study drug randomization:

* < 80% of CGM readings available over the last 2-week period
* Time spent in hypoglycemia (i.e., < 70 mg/dL) for < 5% over a 2-week period on based on CGM reading.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kuei Lin, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amitriptyline: Participants initiated on 25 mg Amitriptyline daily for two weeks during the Titration Period. Amitriptyline dose was increased to 50 mg daily for 8 weeks during the Intervention Period. Finally, the dose of Amitriptyline was reduced to 25 mg daily during the two week Taper Period.
- Placebo: Participants initiated on a daily Placebo capsule matching the 25 mg Amitriptyline during the Titration Period. The daily dose was changed to the Placebo capsule matching the 50 mg Amitriptyline for 8 weeks during the Intervention Period. Finally, the daily dose was changed back to the Placebo matching the 25 mg Amitriptyline during the two week Taper Period.
Period: Overall Study
Arm/Group | Amitriptyline | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Glucose Area Under the Curve (AUC): Values < 70 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The mean AUC for glucose values < 70 mg/dL will be compared between the Amitriptyline and Placebo arms.
Time Frame: 2 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment.
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Glucose Area Under the Curve (AUC): Values < 54 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The mean AUC for glucose values < 54 mg/dL will be compared between the Amitriptyline and Placebo arms.
Time Frame: 2 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Ratio of Self-Reported Hypoglycemic Episodes to Total Hypoglycemic Episodes
Description: Participants will complete a report of all hypoglycemic events experienced during the 2-week surveillance period at the end of the Intervention Phase. The average ratio of self-reported hypoglycemic episodes to total hypoglycemic episodes recorded by Continuous Glucose Monitoring (CGM) will be compared between the Amitriptyline and Placebo arms.
Time Frame: 2 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Total Count of Severe Hypoglycemic Episodes
Description: Severe hypoglycemic episodes, defined by the need from other to administer treatments for hypoglycemia, as reported by patients will be counted and totaled during the Intervention Phase.
Time Frame: 8 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hypoglycemia Episode Count With Blood Glucose < 70 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The number of hypoglycemic episodes for glucose values < 70 mg/dL will be compared between the Amitriptyline and Placebo arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Hypoglycemia Episode Count With Blood Glucose < 54 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The number of hypoglycemic episodes for glucose values < 54 mg/dL will be compared between the Amitriptyline and Placebo arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Average Hypoglycemia Duration With Blood Glucose < 70 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The duration of hypoglycemic episodes for glucose values < 70 mg/dL will be averaged compared between the Amitriptyline and Placebo arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Average Hypoglycemia Duration With Blood Glucose < 54 mg/dL
Description: Continuous Glucose Monitoring (CGM) data will be collected for a 2-week period at the end of the Intervention Phase. The duration of hypoglycemic episodes for glucose values < 54 mg/dL will be averaged compared between the Amitriptyline and Placebo arms.
Time Frame: 2 weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Hypoglycemia Awareness Score by Gold Questionnaire
Description: Participants will complete the Gold questionnaire for hypoglycemia awareness at the baseline and final Intervention Phase visit. The Gold questionnaire is comprised of one question to evaluate the hypoglycemia awareness, with scores from 1 to 7, representing from normal to minimal/no hypoglycemia awareness. The average change in Gold questionnaire score from baseline to end of treatment will be compared between the Amitriptyline and Placebo arms.
Time Frame: 10 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Hypoglycemia Awareness Score by Clarke Questionnaire
Description: Participants will complete the Clarke questionnaire for hypoglycemia awareness at the baseline and final Intervention Phase visit. The Clarke questionnaire is comprised of eight questions to evaluate the hypoglycemia awareness. The answer for each individual question will represent a score (0 or 1). These scores will be summed together to a final score from 0 to 7, representing from normal to minimal/no hypoglycemia awareness. The average change in Clarke questionnaire score from baseline to end of treatment will be compared between the Amitriptyline and Placebo arms.
Time Frame: 10 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Hypoglycemia Awareness Score by Pedersen-Bjergaard Questionnaire
Description: Participants will complete the Pedersen-Bjergaard questionnaire for hypoglycemia awareness at the baseline and final Intervention Phase visit. The Pederson-Bjergaard questionnaire is comprised of one question to evaluate the hypoglycemia awareness, with answers of "Always", "sometimes", "occasionally", "never" or "Do not know". Each answer will represent an awareness status. The change in Pedersen-Bjergaard questionnaire status from baseline to end of treatment will be compared between the Amitriptyline and Placebo arms.
Time Frame: 10 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Hypoglycemia Fear Survey Score
Description: Participants will complete the Hypoglycemia Fear Survey for hypoglycemia fear assessment at the baseline and final Intervention Phase visit. The Hypoglycemia Fear Survey is comprised of 33 questions to evaluate the hypoglycemia awareness. The answer for each individual question will represent a score (0 to 4). These scores will be summed together to a final score from 0 to 132, representing from normal to minimal/no hypoglycemia awareness. The average change in Hypoglycemia Fear Survey questionnaire score from baseline to end of treatment will be compared between the Amitriptyline and Placebo arms.
Time Frame: 10 Weeks
Population: No analysis conducted due to small sample size; study terminated due to low enrollment
Arm/Group | Amitriptyline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 Weeks
Arm/Group | Amitriptyline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amitriptyline (N=1) | Placebo (N=1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT03591458/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT03591458/ICF_001.pdf